CLINICAL TRIAL: NCT06386965
Title: Sevoflurane Versus Propofol: A Comparision on Stress Response in Patients Undergoing Elective Lombar Disc Surgery
Brief Title: Sevoflurane Versus Propofol: Effect on Stress Response
Status: Completed | Type: Observational
Sponsor: Dr. Lutfi Kirdar Kartal Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Merve Bulun Yediyıldız, Anesthesiology Specialist, MD, Dr. Lutfi Kirdar Kartal Training and Research Hospital
Other Study IDs: 010.99/15
Record Dates: First submitted 2024-04-18; First posted 2024-04-26 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Propofol; Sevoflurane; Inflammatory Response
Keywords: propofol; sevoflurane; inflammatory response
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- propofol: General anesthesia will maintain with propofol in this group.
  Interventions: Other: taking blood sample
- sevoflurane: General anesthesia will maintain with sevoflurane in this group.
  Interventions: Other: taking blood sample

INTERVENTIONS:
Other: taking blood sample — A blood sample will be taken from the patients for 3 times to evaluate the stress inflammatory markers.

SUMMARY:
Stress is defined as hormonal and metabolic changes in the biological system that follow any injury. The stress response occurs as a general systemic response to injury and includes a wide range of endocrinological, immunological and hematological effects. The level of stress in the surgical process can affect not only the patients outcome but also the overall health system.

The two main agents used in maintenance for general anesthesia are inhalation and intravenous anesthetics. Both inhalation anesthesia and TIVA (Total Intravenous Anesthesia) approaches provide general anesthesia suitable for surgical operations. However, the mechanisms of action of these two methods differ and are not fully understood.

The aim of investigators' for this study was to investigate the effect of different anesthetic agents on stress inflammatory response in the preoperative, peroperative and postoperative periods.

DETAILED DESCRIPTION:
Lumbar microdiscectomy is the most preferred surgical method in lumbar disc disease and successful results are obtained with the right indication and appropriate surgery. After the operation, rapid and dramatic improvements are observed in terms of pain complaints and neurologic deficits. The recovery process in these patients may be related to many reasons and may also be associated with stress inflammatory marker response.

The two main agents used in maintenance for general anesthesia are inhalation and intravenous anesthetics. Both inhalation anesthesia and TIVA (Total Intravenous Anesthesia) approaches provide general anesthesia suitable for surgical operations.Previous studies have shown that inhalation agents alter immune processes and are proinflammatory. In contrast, propofol has been shown to suppress tumor growth and has anti-inflammatory and antioxidant activities.

The aim of investigators' for this study was to investigate the effect of different anesthetic agents on stress inflammatory response in the preoperative, peroperative and postoperative periods.

This single-center prospective,observational study was approved by Institutional Ethics Committee (Decision number: 2024/010.99/15, Date: 28/02/2024) and was started to performed in accordance with the Declaration of Helsinki. In this study, 40 patients in the ASA I-II group who will be operated electively for lumbar disc herniation between March and June 2023 in the operating room of the Neurosurgery Department of Kartal Dr Lütfi Kırdar City Hospital will be divided into two groups to be maintained with sevoflurane or propofol by appropriate randomization.

Blood samples collected before surgical intervention (T1), intraoperative 30 minutes (T2) and postoperative 12 hours (T3) will be analyzed and parameters that may be related to stress inflammatory response such as glucose, WBC, procalcitonin, CRP, erythrocyte sedimentation rate, transferrin, ferritin, albumin, prealbumin will be compared.

ELIGIBILITY:
Inclusion Criteria:

* Extruded disc
* Motor deficit
* L4-5, L5-S1 levels disc herniation
* 18-65 years
* ASA I-II

Exclusion Criteria:

* Recurrence disc operation
* Narrow channel
* Trauma
* Infection
* Endocrine disease

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Between April and June 2023, ASA I-II, 18-65 years old 40 patients with single level lumbar disc herniation who underwent elective surgery in the neurosurgery operating room were planned to participate.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2024-05-23 (Actual); Primary Completion 2024-06-05 (Actual); Study Completion 2024-06-05 (Actual)

PRIMARY OUTCOMES:
compare inflammatory markers with sevolurane and propofol : glucose, WBC, procalcitonin, CRP, erytrocyte sedimentation rate, ferritin, pre albumin, albumin,tranferrin | preoperative, intraoperative, postoperative 12-24 h (an average of 3 months)
  The primary aim of investigators' for this study was to compare the effect of different anesthetic agents on stress inflammatory response in the preoperative, peroperative and postoperative periods.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Health Science, Kartal Dr Lutfi Kırdar Training and Researh Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Yediyildiz MB, Durmus I, Ak HY, Taskin K, Ceylan MAD, Yuce Y, Cevik B, Aydogmus E. Comparison of inhalation and total intravenous anesthesia on inflammatory markers in microdiscectomy: a double-blind study. BMC Anesthesiol. 2025 May 10;25(1):238. doi: 10.1186/s12871-025-03119-6. PMID 40348954